CLINICAL TRIAL: NCT01072474
Title: Capnography as an Adjunct to Standard Monitoring During Midazolam and Propofol Sedation for ERCP
Brief Title: Capnography During ERCP
Acronym: EndoBreath
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Stefan von Delius, II. Medizinische Klinik der Technischen Universität München
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2680/10
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Hypoxemia; Complications
Keywords: Safety; Sedation; Gastrointestinal endoscopy; Colonoscopy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnography (Experimental): Arm with capnographic monitoring
  Interventions: Procedure: Capnography
- Standard (Placebo Comparator): Standard monitoring.
  Interventions: Procedure: Standard monitoring

INTERVENTIONS:
Procedure: Capnography — Capnographic monitoring
  Arms: Capnography
Procedure: Standard monitoring — Standard monitoring
  Arms: Standard

SUMMARY:
In the study the value of capnography for avoiding complications during sedation for ERCP is evaluated.

DETAILED DESCRIPTION:
In this randomized controlled trial the utility of capnography gets evaluated. Hypoxemia may occur during sedation with midazolam and propofol. Whether hypoxemia may be prevented by an additional capnographic monitoring is subject of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Scheduled for colonoscopy with midazolam and propofol sedation

Exclusion Criteria:

* No informed consent
* ASA V
* Pregnancy
* Prexisting hypotension, bradycardia or hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | From the beginning to the end of the ERCP procedure, i.e. from 0h to approximately 2h

SECONDARY OUTCOMES:
Further complications | From the beginning to the end of the ERCP procedure, i.e. from 0h to approximately 2h

CONTACTS AND LOCATIONS:
Overall Officials: Stefan von Delius, MD, Principal Investigator — Technical University of Munich
Locations (3):
- Germany (3):
  - Technische Universität München, Munich, Bavaria
  - Knappschaftskrankenhaus der Ruhr-Universität Bochum, Bochum
  - Deutsche Klinik für Diagnostik, Wiesbaden

REFERENCES:
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079
- [Derived] Klare P, Reiter J, Meining A, Wagenpfeil S, Kronshage T, Geist C, Heringlake S, Schlag C, Bajbouj M, Schneider G, Schmid RM, Wehrmann T, von Delius S, Riphaus A. Capnographic monitoring of midazolam and propofol sedation during ERCP: a randomized controlled study (EndoBreath Study). Endoscopy. 2016 Jan;48(1):42-50. doi: 10.1055/s-0034-1393117. Epub 2015 Sep 28. PMID 26415090
- See also: II. Medizinische Klinik der Technischen Universität München — http://www.med2.med.tu-muenchen.de/